CLINICAL TRIAL: NCT04000958
Title: Optimized Inhalation Therapy Based on Peak Inspiratory Flow Rates Measured Against the Simulated Resistance in Patients Recovering From Acute Exacerbation of Chronic Obstructive Pulmonary Disease: a Randomized Trial (PIFR-OIT Study)
Brief Title: PIFR-based Inhalation Therapy in Patients Recovering From AECOPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2019-142
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIFR group (Experimental)
  Interventions: Drug: PIRF measured by InCheck DIAL
- control group (Active Comparator)
  Interventions: Drug: Regular treament

INTERVENTIONS:
Drug: PIRF measured by InCheck DIAL — Peak inspiratory flow rates(PIFR) will be measured using the InCheck DIAL(Clement Clarke International Ltd, Harlow, UK and Alliance Tech Medical). The InCheck DIAL is accurate to +/- 10% or 10 L/min, whichever is greater, and can measure flows in the range of 15 to 120 L/min. Dry powder inhaler(DPI) is to be prescribed if PIFRr is over 60L/min, otherwise pressure metered dose inhaler(pMDI) with spacer is given. All the patients will be given inhaled corticosteroid（ICS）/long-acting β agonist（LABA）. For symptomatic patients, long-acting anticholinergic agents(LAMA) will also be used.
  Arms: PIFR group
Drug: Regular treament — The choice of inhalers depends on physician's evaluation. The medication is the same as experimental group.
  Arms: control group

SUMMARY:
This study is designed to determine whether the optimized inhalation therapy based on peak inspiratory flow rates (PIFR) measured against the simulated resistance can reduce the rate of treatment failure in patients recovering from acute exacerbation of chronic obstructive pulmonary disease (AECOPD). Errors in inhaler use and quality of life are also to be evaluated.

The study will recruit 460 patients with AECOPD whose exacerbated symptoms are relieved by 5-7 days of standard therapy. The participants are divided into PIFR group and control group in a 1:1 ratio according to a random number table method. All the patients will be given inhaled corticosteroid（ICS）/long-acting β agonist（LABA） (budesonide/ formoterolSymbicort turbuhaler® 160/4.5 μg bid or Beclometasone/ Formoterol Foster® pressure metered dose inhaler(pMDI) 100/6 μg 2 puff bid). For symptomatic patients before acute exacerbation, Spiriva handihaler® 18μg qd or Spiriva respimat® 2.5μg qd will be prescribed in combination with ICS/LABA. For PIFR group, PIFR is measured by InCheck DIAL(Clement Clarke International Ltd, Harlow, UK and Alliance Tech Medical). If PIFR is less than 60L/min , the patient will be given pMDI with spacer. If PIFR value is over 60 L/min, the patient will be given dry powder inhaler(DPI).). The control group will be given DPI or pMDI with spacer according to the judgment of a respiratory physician. Both groups will be taught to use the device after the prescription, and then be reminded to use medication via a WeChat public account.

The primary endpoint of the study is the 30-day treatment failure including AECOPD recurrence resulting in an emergency visit, admission, or need for intensified medication). The secondary endpoints of the study are the error rate of inhalation device use, satisfaction with inhalation devices, symptoms and quality of life, 30-day mortality, chronic obstructive pulmonary diseases(COPD)-related treatment costs and PIFR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute exacerbation of chronic obstructive pulmonary disease(AECOPD) whose acute respiratory symptoms have been controlled after 5-7 day-standard AECOPD treatment including atomized or inhaled brochodilator plus oral or intravenous glucocorticoid (prednisone equivalent dose 40-50mg) or Pulmicort 2mg atomization Bid plus broad-spectrum antibiotics.
* Patients with moderate and above chronic obstructive pulmonary disease diagnosed by spirometry, ie, forced expiratory volume in one second(FEV1)/forced vital capacity(FVC) <70% post-bronchodilator and FEV1% predicted value <80%.
* Patients have signed an informed consent form.

Exclusion Criteria:

* Patients who is already using home nebulization therapy because of the severity of the illness.
* Patients with bronchial asthma, pulmonary interstitial fibrosis, bronchiectasis, pulmonary embolism and other lung diseases; or hypertension, heart disease, chronic liver and kidney disease, diabetes, chronic gastrointestinal diseases, malignant tumors, critically ill patients.
* Patient's mental state cannot match the observation or suffer from cognitive impairment.
* Patient's peak inspiratory flow rates (PIFR) is less than 20L/min.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
30-day treatment failure rate | 30 days
  Treatment failure means AECOPD recurrence resulting in an emergency visit, admission, or need for intensfied medication.

SECONDARY OUTCOMES:
the error rate of inhalation device use | 30 days/ 90 days
satisfaction with inhalation devices | 30 days/ 90 days
  Patients' satisfaction with inhalation devices will be assessed by the following items. If the patient meets any of the following, the result will be unsatisfactory:
  1. The patient has forgotten to use the inhaler.
  2. The patient has forgotten to use the inhaler in the last two weeks.
  3. The patient has reduced the frequency of using inhaler without medical advice.
  4. The patient has forgotten to bring an inhaler when traveling or leaving home.
  5. The patient has quitted the inhaler without medical advice when feeling his condition improved.
  6. The patient has felt it difficult to comply with the COPD treatment plan.
  7. The patient has felt it difficult to use the inhaler.
score of St.George's Respiratory Questionnaire(SGRQ) | 30 days/ 90 days
  St.George's Respiratory Questionnaire(SGRQ) is used to assess patient's quality of life.
  The SGRQ scale range is from 0 to 100. The higher the score is, the more severe the impact of COPD on patient' life is.
30-day mortality | 30 days
COPD-related treatment costs | 30 days/ 90 days
Peak Inspiratory Flow Rates（PIFR） | 30 days/ 90 days
90-day mortality | 90 days
score of modified British medical research council(mMRC) | 30 days/ 90 days
  Modified British medical research council(mMRC) is used to assess patient's symptoms.
  The mMRC scale range is from 0 to 4. The higher the score is, the more severe the patient's dyspnea is.
score of COPD assessment test(CAT) | 30 days/ 90 days
  COPD assessment test(CAT) is used to assess patient's symptoms. The CAT scale range is from 0 to 40. A score of 0-10 indicates the patient is slightly affected by COPD. A score of 11-20 indicates the patient is moderately affected by COPD. A score of 21-30 indicates the patient is seriously affected by COPD. A score of 31-40 indicates the patient is extremely affected by COPD.

CONTACTS AND LOCATIONS:
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hua J, Zhang W, Cao HF, Du CL, Ma JY, Zuo YH, Zhang J. Effect of PIFR-based optimised inhalation therapy in patients recovering from acute exacerbation of chronic obstructive pulmonary disease: protocol of a prospective, multicentre, superiority, randomised controlled trial. BMJ Open. 2020 May 7;10(5):e034804. doi: 10.1136/bmjopen-2019-034804. PMID 32385061